CLINICAL TRIAL: NCT03165279
Title: ZEnith AlPHa for AneurYsm Repair (ZEPHYR)
Brief Title: ZEnith AlPHa for AneurYsm Repair
Acronym: ZEPHYR
Status: Completed | Type: Observational
Sponsor: Philippe Cuypers (Other)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor-Investigator, Philippe Cuypers, MD, PhD, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Other Study IDs: ZEPHYR
Record Dates: First submitted 2017-05-16; First posted 2017-05-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with AAA: Patient will receive a 'Zenith Alpha Abdominal stentgraft' as intervention to eliminate the abdominal aortic aneurysm.
  Interventions: Procedure: Zenith Alpha Abdominal stentgraft

INTERVENTIONS:
Procedure: Zenith Alpha Abdominal stentgraft

SUMMARY:
To prospectively collect 'real world' performance data on the Zenith AlphaTM Abdominal Endovascular Graft for endovascular aneurysm repair, inside and outside instructions for use. To assess clinical efficacy of the low-profile device to treat patients with abdominal aortic aneurysm (AAA), to assess the use of the new delivery and deployment system of the Zenith AlphaTM Abdominal Endovascular Graft. Primary endpoint is the proportion of subjects who experience successful treatment at 1 year post-implant; defined by technical success and clinical success.

DETAILED DESCRIPTION:
The ZEPHYR registry has two major objectives:

1. to prospectively collect 'real world' safety, durability and clinical performance data on the Zenith AlphaTM Abdominal Endovascular Graft in subjects with infrarenal abdominal aortic or aorto-iliac aneurysms.
2. To increase the clinical evidence about the safety and effectiveness of the Zenith AlphaTM Abdominal Endovascular Graft by creating a database that can be pooled and/or compared with databases available on this and other stent graft systems.

The ZEPHYR registry is a multi-center, post-market, non-randomized, single-arm prospective study. The study has no controls, as it is descriptive in nature. It will recruit approximately 450 subjects from high-volume sites across Germany and the BeNeLux. Study is open to consecutively enrolled subjects (20-50 per site) whou in the opinion of the investigator are candidates for endovascular AAA repair. The sites are recommended to schedule the subject's post-operative follow-up visits based on the current standard care in endovascular aneurysm repair (EVAR) therapy, which is generally at 1 month, 1 year and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or minimum age as required by local regulations
* Non-ruptured AAA with maximum diameter ≥50mm or enlargement >5mm over 6 months and neck length ≥10mm (site-reported)
* Elective EVAR
* Intention to electively implant the Zenith AlphaTM AAA Endovascular Graft
* Signed informed consent form

Exclusion Criteria:

* Intolerance to contrast media
* High probability of non-adherence to physician's follow-up requirements
* Current participation in a concurrent trial which may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with defined AAA who are elegible for surgery
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Successful treatment | 1 year
  Proportion of subjects who experience successful treatment at 1 year post-implant; defined by technical success and clinical success.

SECONDARY OUTCOMES:
Treatment success | 1 month
  Proportion of subjects who experience successful treatment at 1 month post-implant; defined by technical success and clinical success.
Treatment success | 2 years
  Proportion of subjects who experience successful treatment at 2 years post-implant; defined by technical success and clinical success.
All-cause mortality | at 1 month, 1 year and at 2 years
  All-cause mortality
Major adverse events | at 1 month, 1 year and at 2 years
  all-cause mortality, bowel ischemia, myocardial infarction, paraplegia, procedural blood loss >1000 cc, renal failure requiring dialysis, respiratory failure, stroke
Aneurysm related mortality | up to 30 days after index procedure or within 30 days after aneurysm-related reintervention
  death from rupture, device-related death, death within 30 days of index procedure, death within 30 days of any aneurysm-related reintervention
Stent graft migration of >5mm (with 30 days measurement as baseline) | at 1 year and at 2 years
  Stent graft migration of >5mm (with 30 days measurement as baseline)
Endoleak | at initial procedure, 1 month, 1 year and at 2 years
  Any type of endoleak; tabulated by type (Ia, Ib, II or III)
Amount of secondary procedures to correct endoleaks | From the day after the initial procedure up to 2 years after the initail procedure (which is the end of the follow up period for this registry)
  Secondary procedures to correct endoleaks
Amount of secondary procedures for occlusion and/or kinking to restore stent graft function (endovascular and open procedures) | From the day after the initial procedure up to 2 years after the initail procedure which is the end of the follow up period
  Amount of secondary procedures for occlusion/kinking to restore stent graft function (endovascular and open surgical procedures)
Amount of secondary surgical interventions for stent graft infection | From the day after the initial procedure up to 2 years after the initail procedure which is the end of the follow up period
  Amount of secondary surgical intervention for stent graft infection
Amount of major lower limb amputation | From the day after the initial procedure up to 2 years after the initail procedure (which is the end of the follow up period for this registry)
  Amount of major lower limb amputation
Which kind of vascular access is used during surgical intervention | at the primary procedure
  Vascular access can either be unilateral, bilateral, open access or percutaneus access
Access site complications | during procedure up to 45 days
  Hematoma, false aneurysm, vessel injury, primary conversion to femoral cutdown, surgical reintervention postoperative, false aneurysm at puncture site
Amount of secondary open surgical interventions | From the day after the initial procedure up to 2 years after the initail procedure (which is the end of the follow up period of this registry)
  Amount of secondary open surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuypers, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (12):
- Belgium (3):
  - Imelda Hospital, Bonheiden
  - Hospital Oost Limburg, Genk
  - University Hospital Gent, Ghent
- Germany (4):
  - Hospital Frankfurt Höchst, Frankfurt am Main
  - University hospital Hamburg, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Hospital Nürnberg Süd, Nuremberg
- Netherlands (5):
  - Catharina Hospital, Eindhoven, North Brabant
  - VUmc, Amsterdam
  - MUMC+, Maastricht
  - Maasstad Hospital, Rotterdam
  - HagaHospital, The Hague

IPD SHARING:
Plan to Share IPD: No